CLINICAL TRIAL: NCT03712345
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Phase II Efficacy and Safety Study of IFX-1 in Add-On to Standard of Care in Granulomatosis With Polyangiitis (GPA) and Microscopic Polyangiitis (MPA)
Brief Title: Safety and Efficacy Study of IFX-1 in add-on to Standard of Care in GPA and MPA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to COVID-19 pandemic outbreak and its impact on overall study activities. All efforts were made to ensure that participants that were enrolled and/or were still in the study will continue to receive treatment and follow-up until study completion.
Sponsor: InflaRx GmbH (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IFX-1-P2.6
Record Dates: First submitted 2018-10-16; First posted 2018-10-19 (Actual); Results first posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Granulomatosis With Polyangiitis (GPA); Microscopic Polyangiitis (MPA)
Keywords: Granulomatosis with Polyangiitis (GPA); Microscopic Polyangiitis (MPA); IFX-1; ANCA; AAV
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Microscopic Polyangiitis | interventions — vilobelimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- IFX-1 low dose (Experimental): Will receive IFX-1 low dose regimen diluted in sodium chloride solution
  Interventions: Drug: IFX-1 low dose
- IFX-1 high dose (Experimental): Will receive IFX-1 high dose regimen diluted in sodium chloride solution
  Interventions: Drug: IFX-1 high dose
- Placebo (Placebo Comparator): Will receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IFX-1 low dose — Single IV infusions of IFX-1
  Other Names: CaCP29
  Arms: IFX-1 low dose
Drug: IFX-1 high dose — Single IV infusions of IFX-1
  Other Names: CaCP29
  Arms: IFX-1 high dose
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of two dose regimens of IFX-1 as add-on to standard of care (SOC) in subjects with GPA and MPA compared with placebo.

DETAILED DESCRIPTION:
Granulomatosis with polyangiitis (GPA) and microscopic polyangiitis (MPA) are related systemic v anti-neutrophil cytoplasmic antibody (ANCA)-associated vasculitis (AAV), a potentially life-threatening disease.

GPA is a necrotizing vasculitis predominantly involving small- to medium-sized vessels (e.g., capillaries, venules, arterioles, arteries, and veins). MPA is a necrotizing vasculitis that primarily affects capillaries, venules, or arterioles, most commonly manifesting as necrotizing glomerulonephritis and/or pulmonary capillaritis. MPA.

Primed neutrophils are activated by ANCA and generate C5a that engages C5a receptors on neutrophils. Therefore, patients with ANCA-related disease have elevated plasma and urine levels of C5a in active disease and not in remission.

IFX-1 is a monoclonal antibody specifically binding to the soluble human complement split product C5a and the resulting nearly complete blockade of C5a-induced biological effects may be effective in the treatment of subjects with AAV.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥18 years of age.
2. Diagnosis of GPA or MPA according to the definitions of the Chapel Hill Consensus Conference.
3. Have at least one "major" item, or at least three other items, or at least two renal items on the Birmingham Vasculitis Activity Score (BVAS) Version 3.0.
4. New or relapsed GPA or MPA that require treatment with CYC or RTX plus GCs.

Exclusion Criteria:

1. Any other multisystem autoimmune disease
2. Requires mechanical ventilation because of alveolar hemorrhage at Screening.
3. Human immunodeficiency virus, hepatitis B, or hepatitis C viral screening test showing evidence of active or chronic viral infection at Screening or a documented history of the human immunodeficiency virus, hepatitis B, or hepatitis C.
4. Received CYC or RTX 12 weeks before Screening; if on azathioprine (AZA), methotrexate (MTX), mycophenolate mofetil (MMF), or mycophenolate sodium (MPS) at the time of Screening, these drugs must be withdrawn prior to receiving CYC or RTX.
5. Received more than 3 g cumulative high dose intravenous GCs within 4 weeks before Screening.
6. On an oral dose of a GC of more than 10 mg prednisone equivalent at Screening or for more than 6 weeks before Screening.
7. Received a CD20 inhibitor, anti-tumor necrosis factor treatment, abatacept, alemtuzumab, any other experimental or biological therapy, intravenous immunoglobulin or plasma exchange, antithymocyte globulin, or required dialysis within 12 weeks before Screening.
8. Received a live vaccination within 4 weeks before Screening or planned between Screening and Week 24.
9. Female subjects of childbearing potential unwilling or unable to use a highly effective method of contraception (pearl index <1%) such as complete sexual abstinence, combined oral contraceptive, vaginal hormone ring, transdermal contraceptive patch, contraceptive implant, or depot contraceptive injection in combination with a second method of contraception such as condom, cervical cap, or diaphragm with spermicide during the study and for at least 4 weeks after last administration of IFX-1 (timeframes for SOC have to be considered as described in the respective Prescribing Information).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2021-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Korinna Pilz, MD, MS, Study Director — InflaRx GmbH; Peter A. Merkel, MD, MPH, Principal Investigator — University of Pennsylvania
Locations (38):
- United States (33):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Loma Linda University Clinical Trial Center, Loma Linda, California
  - Science Connections, LLC, Doral, Florida
  - University of Miami, Miami, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - LSU Health Sciences Center Shreveport, Shreveport, Louisiana
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University Of MI Medcl Ctr-RHU, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - Northwell Health, LLC PRIME, New Hyde Park, New York
  - Hospital for Special Surgery, New York, New York
  - University of Rochester Medical Center - Strong Memorial Hospital, Rochester, New York
  - UNC Kidney Center, UNC-CH Division of Nephrology and Hypertension, Chapel Hill, North Carolina
  - Trinity Medical Group, Minot, North Dakota
  - Ohio State University Clinical Trials Management Office, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - BRCR Medical Center, Inc., Camp Hill, Pennsylvania
  - Altoona Center for Clinical Research, P.C., Duncansville, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Low Country Rheumatology, PA, North Charleston, South Carolina
  - Adriana Pop Moody Clinic PA, Corpus Christi, Texas
  - Texas Health Resources, Dallas, Texas
  - Texas Research Institute, Fort Worth, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - UVA University Physicians Charlottesville, Charlottesville, Virginia
  - West Virginia University, Morgantown, West Virginia
- Canada (5):
  - University of Alberta Hospital, Edmonton, Alberta
  - St. Josephs Healthcare, Hamilton, Ontaria
  - Mount Sinai Hospital, Toronto, Ontario
  - CHUM Centre de Recherche, Québec, Quebec
  - Centre de Recherche Musculo-Squelettique, Trois-Rivières, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Serling-Boyd N, Wallace ZS. Management of primary vasculitides with biologic and novel small molecule medications. Curr Opin Rheumatol. 2021 Jan;33(1):8-14. doi: 10.1097/BOR.0000000000000756. PMID 33164993

RESULTS

PARTICIPANT FLOW:
Groups:
- IFX-1 High Dose: Will receive IFX-1 high dose regimen diluted in sodium chloride solution
  IFX-1: Single IV infusions of IFX-1
- IFX-1 Low Dose: Will receive IFX-1 low dose regimen diluted in sodium chloride solution
  IFX-1: Single IV infusions of IFX-1
Period: Overall Study
Arm/Group | IFX-1 High Dose | IFX-1 Low Dose | Placebo
Started | 6 | 7 | 7 (One participant was mistakenly randomized, but never treated because the participant was a screening failure.)
Completed | 6 | 7 | 6
Not Completed | 0 | 0 | 1
Not completed — Failure to meet randomization criteria | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | IFX-1 Low Dose | IFX-1 High Dose | Placebo | Total
Number analyzed (Participants) | 7 | 6 | 6 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (15.1) | 54.8 (12.0) | 56.5 (16.2) | 59.1 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 3 | 13
  Male | 2 | 1 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 4
  Not Hispanic or Latino | 6 | 4 | 5 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 5 | 5 | 14
  Asian | 1 | 0 | 0 | 1
  Multiple | 1 | 0 | 0 | 1
  Other | 1 | 1 | 1 | 3
AAV disease type [Count of Participants; unit: Participants]
  GPA | 5 | 4 | 4 | 13
  MPA | 2 | 2 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Participants With at Least One TEAE Per Treatment Group.
Description: Number and percentage of participants who experience at least one treatment-emergent adverse event (TEAE) per treatment group.
Time Frame: Week 24
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | IFX-1 High Dose | IFX-1 Low Dose | Placebo
Number analyzed (Participants) | 6 | 7 | 6
Participants | 6 | 7 | 5

2. Secondary Outcome: Percentage of Participants Achieving Clinical Response
Description: Efficacy Endpoint based on clinical response evaluated through BVAS. Clinical response is defined as a reduction in BVAS of ≥50% and no worsening in any body system and no administration of rescue medication prior to the response assessment.
Time Frame: Week 16
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | IFX-1 High Dose | IFX-1 Low Dose | Placebo
Number analyzed (Participants) | 5 | 7 | 6
Participants | 5 | 6 | 6

3. Secondary Outcome: Percentage of Participants With Clinical Remission (BVAS = 0)
Description: Efficacy Endpoint that evaluates participants with complete remission
Time Frame: Week 16
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | IFX-1 High Dose | IFX-1 Low Dose | Placebo
Number analyzed (Participants) | 5 | 7 | 6
Participants | 3 | 6 | 4

4. Secondary Outcome: IFX-1 Concentration Pre-dose
Description: Assess the pharmacokinetic of the investigational medicinal product.
Time Frame: Week 16
Population: Safety Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | IFX-1 High Dose | IFX-1 Low Dose | Placebo
Number analyzed (Participants) | 3 | 2 | 6
ng/mL | 115598.80 (82.84) | 7258.96 (45.57) | 38.09 (137.68)

5. Secondary Outcome: IFX 1 Concentration at Predose (0 Hours), After the End of the Infusion (+10minutes), and at 2, 6, 24, and 48 Hours After the Start of the Infusion for Participants in the PK Substudy
Description: Analyze the IMP plasma concentration using a PK model: IFX 1 concentration at predose (0 hours), after the end of the infusion (+10minutes), and at 2, 6, 24, and 48 hours after the start of the infusion for participants in the PK substudy
Time Frame: Weeks 1, 4 and 16
Population: Safety Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | IFX-1 High Dose | IFX-1 Low Dose | Placebo
Number analyzed (Participants) | 6 | 7 | 6
ng/mL | NA (NA) — Due to early termination of the study, the PK substudy did not enroll the planned number of 15 participants. Only one of the participants randomized to treatment other than Placebo gave initial consent and did not withdraw consent for the PK substudy at a later timepoint, such that the planned analysis could not be performed but data was only listed. | NA (NA) — Due to early termination of the study, the PK substudy did not enroll the planned number of 15 participants. Only one of the participants randomized to treatment other than Placebo gave initial consent and did not withdraw consent for the PK substudy at a later timepoint, such that the planned analysis could not be performed but data was only listed. | NA (NA) — Due to early termination of the study, the PK substudy did not enroll the planned number of 15 participants. Only one of the participants randomized to treatment other than Placebo gave initial consent and did not withdraw consent for the PK substudy at a later timepoint, such that the planned analysis could not be performed but data was only listed.

6. Secondary Outcome: C5a Plasma Concentration
Description: Pharmacodynamic parameter concentration
Time Frame: Week 16
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | IFX-1 High Dose | IFX-1 Low Dose | Placebo
Number analyzed (Participants) | 4 | 3 | 6
ng/mL | 9.4475 (7.9414) | 37.1361 (9.7106) | 31.6571 (6.9818)

7. Secondary Outcome: IFX-1 Blocking Activity 2.5 nM
Description: Pharmacodynamic Parameter of IFX-1 blocking activity 2.5 nM
Time Frame: Week 16
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: percentage of IFX-1 blocking activity
Arm/Group | IFX-1 High Dose | IFX-1 Low Dose | Placebo
Number analyzed (Participants) | 3 | 3 | 0
percentage of IFX-1 blocking activity | 103.873 (4.667) | 82.383 (21.957) |

8. Secondary Outcome: IFX-1 Blocking Activity 10 nM
Description: Pharmacodynamic Parameter of IFX-1 blocking activity 10 nM
Time Frame: Week 16
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: percentage of IFX-1 blocking activity
Arm/Group | IFX-1 High Dose | IFX-1 Low Dose | Placebo
Number analyzed (Participants) | 3 | 3 | 0
percentage of IFX-1 blocking activity | 101.693 (0.771) | 60.473 (29.531) |

ADVERSE EVENTS:
Time Frame: 26 weeks
Arm/Group | IFX-1 High Dose | IFX-1 Low Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 2/6 | 1/7 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 7/7 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IFX-1 High Dose (N=6) | IFX-1 Low Dose (N=7) | Placebo (N=6)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IFX-1 High Dose (N=6) | IFX-1 Low Dose (N=7) | Placebo (N=6)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal rigidity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral lichen planus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Weight increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood immunoglobulin G (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal paraesthesia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 2 (2) | 1 (1)
Night blindness (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Scleritis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Steroid diabetes (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Anhedonia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 0 (0)
Vulvovaginal rash (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/45/NCT03712345/Prot_SAP_000.pdf